CLINICAL TRIAL: NCT04334096
Title: Long-term Improvement of Quality of Life in Breast Cancer Patients With Tailored Quality of Life Diagnosis and Therapy: Implementation Into Routine Care
Brief Title: Long-term Improvement of Quality of Life in Breast Cancer Patients With Quality of Life Diagnosis and Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tumor Center Regensburg (Other)
Collaborators: German Cancer Aid (Other)
Responsible Party: Principal Investigator, Prof. Dr. Monika Klinkhammer-Schalke, Director of the Tumor Center Regensburg, Tumor Center Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TUZ-QL-Mamma-16; 111169 (Other Grant/Funding Number: German Cancer Aid)
Record Dates: First submitted 2020-03-26; First posted 2020-04-06 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Quality of Life; Breast Cancer; Breast Neoplasms
Keywords: quality of life; breast cancer; complex intervention; long-term implementation; health services research
MeSH Terms: conditions — Breast Neoplasms | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QoL diagnosis and therapy (Experimental): The first quality of life (QoL) measurement is conducted in the hospital after surgery via a digital questionnaire (EORTC QLQ-C30, QLQ-BR23) on a tablet computer. Further QoL measures are accomplished via paper-pencil in the practice of the patient's physician during aftercare (3, 6, 9, 12, 18, 24 months after surgery). Paper questionnaires are transferred by fax to a local server, automatically processed, digitized and stored in a database, and transferred back to the physician's practice (email or fax depending on preference) in form of a QoL profile. The immediate response enables patient and physician to discuss the QoL profile right away. Specific therapeutic options for the treatment of QoL have been defined: psychotherapy, social counseling, pain therapy, physiotherapy, nutrition counseling, fitness. To provide continuous medical education, quality circles for each therapeutic option have been founded. Physicians receive a list with addresses of all quality circle members.
  Interventions: Behavioral: quality of life pathway

INTERVENTIONS:
Behavioral: quality of life pathway — The first quality of life (QoL) measurement is conducted in the hospital after surgery via a digital questionnaire (EORTC QLQ-C30, QLQ-BR23) on a tablet computer. Further QoL measures are accomplished via paper-pencil in the practice of the patient's physician during aftercare (3, 6, 9, 12, 18, 24 months after surgery). Paper questionnaires are transferred by fax to a local server, automatically processed, digitized and stored in a database, and transferred back to the physician's practice (email or fax depending on preference) in form of a QoL profile. The immediate response enables patient and physician to discuss the QoL profile right away. Specific therapeutic options for the treatment of QoL have been defined: psychotherapy, social counseling, pain therapy, physiotherapy, nutrition counseling, fitness. To provide continuous medical education, quality circles for each therapeutic option have been founded. Physicians receive a list with addresses of all quality circle members.
  Other Names: quality of life diagnosis and therapy; quality of life pathway

SUMMARY:
The purpose of the study is the long-term implementation of a system with quality of life diagnosis and tailored therapeutic options in order to improve quality of life of patients with breast cancer during follow-up.

DETAILED DESCRIPTION:
The implementation of quality of life (QoL) concepts in routine care is still an open matter. A pathway with QoL diagnosis and therapeutic options for patients with breast cancer and colorectal cancer has been designed, implemented, and evaluated as guided by the Medical Research Council framework for developing and testing complex interventions. It could be demonstrated that patients with breast cancer and colorectal cancer profited from the diagnosis of QoL deficits and tailored therapeutic options in their treatment.

The next step is the long-term implementation of the QoL pathway into routine care. In a prospective, single-arm study 200 patients with breast cancer are planned to be recruited. QoL is measured (EORTC QLQ-C30, QLQ-BR23) after surgery (baseline) and during aftercare (3, 6, 9, 12, 18, 24 months). Results of QoL measurements are automatically processed via an electronic data processing (EDP)-aided system and are directly presented to the coordinating practitioner (physician who cares for the patient during aftercare) and the patient in a QoL profile that can be discussed during the current medical appointment. The profile consists of eleven dimensions on scales of 0-100. A cutoff score <50 points defines a need for QoL therapy. Specific therapeutic options for the treatment of QoL have been identified: psychotherapy, social counseling, pain therapy, physiotherapy, nutrition counseling, and fitness. To provide continuous medical education, quality circles for each therapy option have been founded. Coordinating practitioners receive a list with addresses of all quality circle members.

The primary endpoint of the study is the proportion of patients with a need for QoL therapy 6 months after surgery as well as the evaluation of clinical relevance of the QoL pathway by patients and physicians.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer
* operated in one of two participating certified centers for breast cancer (Caritas-Krankenhaus St. Josef, Klinik für Frauenheilkunde und Geburtshilfe, Regensburg; Krankenhaus Barmherzige Brüder, Klinik St. Hedwig, Poliklinik für Frauenheilkunde und Geburtshilfe, Regensburg)
* informed consent

Exclusion Criteria:

* unavailability of recruiting study clinician
* patient misclassified in the operation schedule (no breast neoplasm)
* coordinating practitioner refused trial participation
* no "Nachsorgekalendernummer" available ("Nachsorgekalendernummer": unique number of the diary the patient receives in the hospital for aftercare during breast cancer)
* patient from district outside the defined study region
* age under 18 years
* pregnancy
* patient unable to fill out the QoL questionnaire (physical, psychological, cognitive, language reasons)
* patient refused trial participation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2019-01-18 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
proportion of patients with a need for QoL therapy | 6 months after the date of surgery for breast cancer
  a need for QoL therapy is defined as a score <50 points in at least one of eleven QoL dimensions of the EORTC QLQ-C30 and QLQ-BR23 (scales: global quality of life, physical, role, emotional, cognitive, social functioning, pain, fatigue, financial situation, body image, arm symptoms); scores in each dimension are uniformly transformed to dimensions ranging from 0 to 100, with 0 denoting the negative (low functioning, high symptom burden) and 100 the positive end (high functioning, low symptom burden) of the continuum.

SECONDARY OUTCOMES:
proportions of patients with a need for QoL therapy in each dimension of the QoL profile | 3, 6, 9, 12, 18, and 24 months after the date of surgery for breast cancer
  a need for QoL therapy is defined as a score <50 points on each single QoL dimension of the EORTC QLQ-C30 and QLQ-BR23 (scales: global quality of life, physical, role, emotional, cognitive, social functioning, pain, fatigue, financial situation, body image, arm symptoms); scores in each dimension are uniformly transformed to dimensions ranging from 0 to 100, with 0 denoting the negative (low functioning, high symptom burden) and 100 the positive end (high functioning, low symptom burden) of the continuum.
patient evaluation | 6 and 24 months after the date of surgery for breast cancer
  semistructured, self-created questionnaire composed of quantitative and qualitative questions to evaluate clinical relevance of the QoL pathway for patients; for each single question answers are analyzed dichotomously (yes/no) and reported as absolute and relative frequencies
physician evaluation | 6 and 24 months after the date of surgery for breast cancer
  semistructured, self-created questionnaire composed of quantitative and qualitative questions to evaluate clinical relevance of the QoL pathway for physicians; for each single question answers are analyzed dichotomously (yes/no) and reported as absolute and relative frequencies

CONTACTS AND LOCATIONS:
Overall Officials: Monika Klinkhammer-Schalke, MD, Prof., Study Chair — Tumor Center Regensburg; Patricia Lindberg-Scharf, PhD, Principal Investigator — Tumor Center Regensburg; Brunhilde Steinger, MD, Principal Investigator — Tumor Center Regensburg
Locations (1):
- Tumor Center Regensburg, Institute of Quality Management and Health Services Research of the University of Regensburg, Regensburg, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized IPD that underlie the results in a publication are planned to be made available upon request of scientists.
Supporting Information: Study Protocol
Time Frame: 6 months after date of publication until 60 months after date of publication
Access Criteria: Data will be made available to other scientists upon request for nonprofit research. The contact address is monika.klinkhammer-schalke@ukr.de. Scientists are required to send their predefined statistical analysis plan. Together with the scientific review board of the Tumor Center Regensburg a decision will be made based on the quality and usefulness of planned statistical analysis. In case of a positive decision the scientist is required to sign a contract for data usage before receiving anonymized IPD.

REFERENCES:
- [Background] Klinkhammer-Schalke M, Steinger B, Koller M, Zeman F, Furst A, Gumpp J, Obermaier R, Piso P, Lindberg-Scharf P; Regensburg QoL Study Group. Diagnosing deficits in quality of life and providing tailored therapeutic options: Results of a randomised trial in 220 patients with colorectal cancer. Eur J Cancer. 2020 May;130:102-113. doi: 10.1016/j.ejca.2020.01.025. Epub 2020 Mar 13. PMID 32179445
- [Background] Klinkhammer-Schalke M, Lindberg P, Koller M, Wyatt JC, Hofstadter F, Lorenz W, Steinger B. Direct improvement of quality of life in colorectal cancer patients using a tailored pathway with quality of life diagnosis and therapy (DIQOL): study protocol for a randomised controlled trial. Trials. 2015 Oct 14;16:460. doi: 10.1186/s13063-015-0972-y. PMID 26467994
- [Background] Klinkhammer-Schalke M, Koller M, Steinger B, Ehret C, Ernst B, Wyatt JC, Hofstadter F, Lorenz W; Regensburg QoL Study Group. Direct improvement of quality of life using a tailored quality of life diagnosis and therapy pathway: randomised trial in 200 women with breast cancer. Br J Cancer. 2012 Feb 28;106(5):826-38. doi: 10.1038/bjc.2012.4. Epub 2012 Feb 7. PMID 22315052
- [Background] Klinkhammer-Schalke M, Koller M, Ehret C, Steinger B, Ernst B, Wyatt JC, Hofstadter F, Lorenz W; Regensburg QoL Study Group. Implementing a system of quality-of-life diagnosis and therapy for breast cancer patients: results of an exploratory trial as a prerequisite for a subsequent RCT. Br J Cancer. 2008 Aug 5;99(3):415-22. doi: 10.1038/sj.bjc.6604505. PMID 18665187
- [Background] Klinkhammer-Schalke M, Koller M, Wyatt JC, Steinger B, Ehret C, Ernst B, Hofstadter F, Lorenz W. Quality of life diagnosis and therapy as complex intervention for improvement of health in breast cancer patients: delineating the conceptual, methodological, and logistic requirements (modeling). Langenbecks Arch Surg. 2008 Jan;393(1):1-12. doi: 10.1007/s00423-007-0210-5. Epub 2007 Jul 28. PMID 17661076
- [Derived] Lindberg-Scharf P, Steinger B, Koller M, Hofstadter A, Ortmann O, Kurz J, Sasse J, Klinkhammer-Schalke M. Long-term improvement of quality of life in patients with breast cancer: supporting patient-physician communication by an electronic tool for inpatient and outpatient care. Support Care Cancer. 2021 Dec;29(12):7865-7875. doi: 10.1007/s00520-021-06270-1. Epub 2021 Jun 27. PMID 34176020